CLINICAL TRIAL: NCT02699203
Title: Detection of Salivary Insulin Following Low Versus High Carbohydrate Meals in Humans
Brief Title: Detection of Salivary Insulin Following Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H15-02638
Record Dates: First submitted 2016-02-22; First posted 2016-03-04 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2016-02

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-carbohydrate meal (Experimental): High carbohydrate breakfast meal consisting of oatmeal and berries.
  Interventions: Behavioral: High-carbohydrate meal
- Low-carbohydrate meal (Experimental): Low carbohydrate breakfast meal consisting of eggs and avocado.
  Interventions: Behavioral: Low-carbohydrate meal

INTERVENTIONS:
Behavioral: High-carbohydrate meal — Participants will consume a high-carbohydrate low fat meal. The macronutrients content will be 55% carbohydrate, 25% protein and 20% fat providing 400-500 kcal. Between interventions there will be at least a 48-hours washout, where participants are encouraged to return to their baseline dietary habits.
  Arms: High-carbohydrate meal
Behavioral: Low-carbohydrate meal — Participants will consume a low-carbohydrate high fat meal. The macronutrients content will be 10% carbohydrate, 25% protein and 65% fat and will provide 400-500 kcal (matched to the high carbohydrate meal). Between interventions there will be at least a 48-hours washout, where participants are encouraged to return to their baseline dietary habits.
  Arms: Low-carbohydrate meal

SUMMARY:
In addition to its role as the major regulator of glucose uptake into peripheral tissues, the hormone insulin is also a primary regulator of fat storage and fat burning of the body. Mechanistic animal studies have shown that high insulin may be the initial trigger for weight gain and be the proximal cause of obesity. There is currently no quick or non-invasive way of measuring insulin as research and clinical techniques require collection of a blood sample followed by a complicated and costly biochemical assay. The investigators will test the hypothesis that insulin levels can be accurately measured in saliva in humans following meals that elicit high and low blood insulin responses. Findings will help determine if insulin can be use as a valid fluid to track insulin changes in humans.

DETAILED DESCRIPTION:
Lean and obese healthy participants will consume both a high carbohydrate meal and a low carbohydrate meal designed to elicit different insulin responses on two separate occasions. Blood samples and saliva samples will be collected for 2 hours following each meal and insulin will be measured in both plasma and saliva. The relationship between plasma and saliva insulin following the two meals will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.5-24.9 or over 30.0 kg/m2

Exclusion Criteria:

* Diabetes or other medical conditions affecting glucose or insulin levels
* Smoker
* Competitive athlete
* Vegan or vegetarian

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Peak plasma insulin level | 0-120 minutes
  Peak plasma insulin concentration in high carbohydrate versus low carbohydrate arm.

SECONDARY OUTCOMES:
Plasma insulin area under the curve | 0-120 minutes
  Area under the curve for plasma insulin in high carbohydrate versus low carbohydrate arm.
Relationship between peak saliva and peak plasma insulin | 0-120 minutes
  Correlation of peak plasma and peak saliva insulin in high carbohydrate versus low carbohydrate arm.
Timing of peak saliva and peak plasma insulin | 0-120 minutes
  Timing of peak plasma and peak saliva insulin in high carbohydrate versus low carbohydrate arm.
Relationship between saliva insulin area under the curve and plasma insulin area under the curve | 0-120 minutes
  Correlation between area under the curve for plasma and saliva insulin in high carbohydrate versus low carbohydrate arm.
Peak saliva insulin level | 0-120 minutes
  Peak salivary insulin in high carbohydrate versus low carbohydrate arm
Saliva insulin area under the curve | 0-120 minutes
  Area under the curve for salivary insulin in high carbohydrate versus low carbohydrate arm

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Little, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No